CLINICAL TRIAL: NCT03142126
Title: Angioseal Groin Management After Left Heart Catheterization
Brief Title: Accelerated Ambulation After Vascular Access Closure Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Providence Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 548976
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2017-05

CONDITIONS: Coronary Angiography; Heart Catheterization
MeSH Terms: interventions — Early Ambulation

STUDY DESIGN:
Intervention Model Description: Eligible patients will receive early ambulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Early Ambulation (Experimental): To affirm the safety and efficacy of ambulation of 20 minutes after diagnostic left heart catheterization.
  Interventions: Device: Early ambulation with Angioseal closure device

INTERVENTIONS:
Device: Early ambulation with Angioseal closure device — To reaffirm safety and efficacy of using Angioseal for early ambulation by patients after femoral artery arteriotomy
  Other Names: Angioseal

SUMMARY:
The researchers are seeking to study whether or not there is benefit in keeping patients flat after Angioseal for extended periods of time after diagnostic heart catheterization or if a more aggressive approach of early ambulation would be just as safe while improving cost and patient comfort.

DETAILED DESCRIPTION:
Diagnostic left heart catheterization is the gold standard to assess coronary anatomy. A number of post procedure closure devices have been used in order to be able to ambulate patients after the procedure. Without closure device of the arterial sheath the typical time a patient must lay flat following a diagnostic left heart catheterization at Providence hospital is approximately six hours. This extended time of having to lie flat for the patient is both uncomfortable and time consuming for hospital employees.

The Angioseal closure device is a vascular plug that has been approved by the FDA in order to seal the femoral artery arteriotomy and allow for a faster ambulation time after cardiac catheterization. Currently, the Angioseal device has been approved for ambulation times of 20 minutes after diagnostic left heart catheterization but a more conservative approach is typically used after device. A very common strategy after Angioseal is to keep the patient flat for 2 hours prior to ambulation and then to keep the patient another hour after ambulation for observation of the femoral site.

While a conservative strategy may be considered safer to the operator the Angioseal device has already been approved for an early ambulation strategy. The goal of this study is to reaffirm the safety and efficacy of using Angioseal for early ambulation. If early ambulation is performed it could improve patient comfort and even reduce cost.

ELIGIBILITY:
Inclusion Criteria: Patients undergoing diagnostic left heart catheterization.

Exclusion Criteria: Patients who do not meet criteria for Angioseal closure after diagnostic left heart catheterization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-08-06 (Actual); Primary Completion 2015-08-05 (Actual); Study Completion 2015-09-05 (Actual)

PRIMARY OUTCOMES:
Failure of device to achieve hemostasis | 20 minutes after procedure
  Continued bleeding after deployment prior to discharge

SECONDARY OUTCOMES:
Pseudoaneurysm | 7-10 days after discharge
  Clinical assessment in office follow-up visit
Groin hematoma | 7-10 days after discharge
  Clinical assessment in office follow-up visit, 7-10 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marcel E Zughaib, MD, Study Director — Program Director-Physician Residency

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romagnoli E, Biondi-Zoccai G, Sciahbasi A, Politi L, Rigattieri S, Pendenza G, Summaria F, Patrizi R, Borghi A, Di Russo C, Moretti C, Agostoni P, Loschiavo P, Lioy E, Sheiban I, Sangiorgi G. Radial versus femoral randomized investigation in ST-segment elevation acute coronary syndrome: the RIFLE-STEACS (Radial Versus Femoral Randomized Investigation in ST-Elevation Acute Coronary Syndrome) study. J Am Coll Cardiol. 2012 Dec 18;60(24):2481-9. doi: 10.1016/j.jacc.2012.06.017. Epub 2012 Aug 1. PMID 22858390
- [Background] Jolly SS, Yusuf S, Cairns J, Niemela K, Xavier D, Widimsky P, Budaj A, Niemela M, Valentin V, Lewis BS, Avezum A, Steg PG, Rao SV, Gao P, Afzal R, Joyner CD, Chrolavicius S, Mehta SR; RIVAL trial group. Radial versus femoral access for coronary angiography and intervention in patients with acute coronary syndromes (RIVAL): a randomised, parallel group, multicentre trial. Lancet. 2011 Apr 23;377(9775):1409-20. doi: 10.1016/S0140-6736(11)60404-2. Epub 2011 Apr 4. PMID 21470671
- [Derived] Brancheau D, Sarsam S, Assaad M, Zughaib M. Accelerated ambulation after vascular access closure device. Ther Adv Cardiovasc Dis. 2018 May;12(5):141-144. doi: 10.1177/1753944718756604. Epub 2018 Feb 8. PMID 29421959